CLINICAL TRIAL: NCT02807662
Title: Meeting the Needs of Pregnant Women With PTSD in Prenatal Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Linda Weinreb, Principal Investigator, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1 R40MC23633-01-00
Record Dates: First submitted 2016-06-14; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; prenatal care
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Intervention mothers receive adapted Seeking Safety intervention delivered by prenatal care advocate over 8 sessions
  Interventions: Behavioral: Adapted Seeking Safety Intervention
- No intervention (No Intervention): Treatment as usual mothers receive usual services of a prenatal care advocate

INTERVENTIONS:
Behavioral: Adapted Seeking Safety Intervention — Intervention participants received Seeking Safety psychosocial education Intervention adapted for prenatal care setting.
  Arms: Experimental

SUMMARY:
The objectives of this research study are to screen 750 pregnant women at risk of trauma-related stress symptoms, and adapt and test an evidence-based intervention for pregnant women with PTSD and sub-threshold PTSD symptoms served by two public payer community health centers.

DETAILED DESCRIPTION:
Studies of Posttraumatic Stress Disorder (PTSD) in pregnant women in public payer settings have shown rates 5 or more times that of other populations, and rates as high as 33% of lifetime PTSD sub-threshold symptoms. PTSD during pregnancy has been linked to poor prenatal care and high risk behaviors such as drug and alcohol use and smoking. Further, PTSD may pose a barrier to care as obstetric procedures and pregnancy may trigger PTSD symptoms and avoidance of care. PTSD is also associated with pregnancy and birth complications and negative postpartum outcomes including excessive weight gain, preterm birth, low birth weight, risk for parenting problems, and increased barriers to breastfeeding. However, screening, identification, and support for PTSD is lacking. This study will screen 750 pregnant women at risk of trauma-related stress symptoms, and adapt and test an evidence-based intervention for pregnant women with PTSD and sub-threshold PTSD symptoms served by two public payer community health centers.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are receiving prenatal care
* 18 years or older
* In the first 20 weeks of pregnancy
* Screen positive for posttraumatic stress disorder

Exclusion Criteria:

* Not pregnant
* Not currently psychotic
* No current suicidal ideation
* Language other than English, Spanish, Vietnamese, and Portuguese

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in posttraumatic stress disorder symptoms | The primary endpoint is one month postpartum
Preterm labor | the primary endpoint is one month postpartum
Birthweight | the primary endpoint is one month postpartum

SECONDARY OUTCOMES:
Number of visits for prenatal care | the primary end point is one month postpartum
Change in depression symptoms | the primary endpoint is one month postpartum
change in coping strategies inventory | the primary endpoint is one month postpartum

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219
- [Derived] Weinreb L, Wenz-Gross M, Upshur C. Postpartum outcomes of a pilot prenatal care-based psychosocial intervention for PTSD during pregnancy. Arch Womens Ment Health. 2018 Jun;21(3):299-312. doi: 10.1007/s00737-017-0794-x. Epub 2017 Nov 7. PMID 29116416